CLINICAL TRIAL: NCT00000237
Title: Buprenorphine Detoxification - BBDVI
Brief Title: Buprenorphine Detoxification - BBDVI - 19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Vermont (Other)
Purpose: Treatment
Other Study IDs: NIDA-06969-19; R01-06969-19
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2005-08-17 (Estimated); Status verified 1997-05

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to examine the long-term efficacy of alternate-day dosing schedules in promoting treatment compliance in the absence of confounding behavioral contingencies.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 1997-05

PRIMARY OUTCOMES:
Drug use
Retention
Weeks abstinent
Weeks continuous abstinence
Overall treatment outcome
Opioid dependence and psychiatric status

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Treatment Research Center, Burlington, Vermont, United States